CLINICAL TRIAL: NCT00003402
Title: Autologous Transplantation With and High Dose BCNU and Melphalan Followed by Consolidation With DCEP Plus Taxol/Cisplatin in Patients With Poor Prognosis Low Grade Non-Hodgkin's Lymphoma and Chronic Lymphocyte Leukemia, Who Have Received < or = 12 Months of Standard Therapy
Brief Title: Peripheral Stem Cell Transplantation Plus Combination Chemotherapy in Treating Patients With Low-Grade Non-Hodgkin's Lymphoma or Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: University of Maryland Greenebaum Cancer Center (Other)
Responsible Party: UM Greenebaum Cancer Center
Purpose: Treatment
Other Study IDs: CDR0000066407; MSGCC-9734; NCI-V98-1439
Record Dates: First submitted 1999-11-01; First posted 2004-03-31 (Estimated); Last update posted 2019-10-17 (Actual); Status verified 2019-10

CONDITIONS: Leukemia; Lymphoma
Keywords: Waldenstrom macroglobulinemia; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; refractory chronic lymphocytic leukemia; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; stage III mantle cell lymphoma; stage IV mantle cell lymphoma; recurrent mantle cell lymphoma
MeSH Terms: conditions — Leukemia; Lymphoma; Waldenstrom Macroglobulinemia; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Follicular; Lymphoma, Mantle-Cell | interventions — Carmustine; Cisplatin; Cyclophosphamide; Dexamethasone; Etoposide; Melphalan; Paclitaxel; Peripheral Blood Stem Cell Transplantation

INTERVENTIONS:
Drug: carmustine
Drug: cisplatin
Drug: cyclophosphamide
Drug: dexamethasone
Drug: etoposide
Drug: melphalan
Drug: paclitaxel
Procedure: bone marrow ablation with stem cell support
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining chemotherapy with peripheral stem cell transplantation may allow the doctor to give higher doses of chemotherapy drugs and kill more cancer cells.

PURPOSE: Phase II trial to study the effectiveness of peripheral stem cell transplantation plus combination chemotherapy in treating patients who have low-grade non-Hodgkin's lymphoma or chronic lymphocytic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the complete and partial response rates to treatment with peripheral blood stem cell supported high dose carmustine and melphalan followed by consolidation therapy with dexamethasone/cyclophosphamide/etoposide/cisplatin (DCEP) and dexamethasone, paclitaxel, and cisplatin in patients with poor prognosis low grade non-Hodgkin's lymphoma or chronic lymphocytic leukemia and no greater than 12 months of prior standard therapy. II. Evaluate the incidence of early deaths (less than 60 days posttransplant) in comparison with historical experience in this patient population. III. Evaluate the toxicity of posttransplantation chemotherapy with DCEP and dexamethasone, paclitaxel, and cisplatin in these patients.

OUTLINE: Patients receive carmustine IV over 2 hours on day -2 and melphalan IV on day -1 followed by peripheral blood stem cell infusion on day 0. At 3 months and 9 months after completion of autologous transplantation, patients receive cyclophosphamide, etoposide, and cisplatin by continuous IV infusion for 4 days plus dexamethasone orally every day for 4 days. At 6 and 12 months after completion of autologous transplantation, patients receive dexamethasone orally every day for 4 days, paclitaxel continuous IV infusion over 6 hours on day 2, and cisplatin continuous IV infusion over 24 hours on day 3.

PROJECTED ACCRUAL: There will be 12-35 patients accrued into this study over 1-2.5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed low grade follicular lymphoma, mantle cell lymphoma, or chronic lymphocytic leukemia with no greater than 12 months of prior standard therapy Follicular lymphoma Must have poor prognosis disease defined as any of the following: Any nodal or extranodal tumor mass with a diameter more than 7 cm Involvement of at least 3 nodal sites, each of which has a diameter greater than 3 cm Systemic symptoms Substantial splenic involvement no greater than 5 cm below left costal margin Serous effusions (ascites, pleural or pericardial effusions) Orbital or epidural involvement Ureteral compression Leukemia presentation (at least 500/microliter) Increased LDH level Greater than 20% bone marrow involvement Mantle cell lymphoma No mantle zone morphology Chronic lymphocytic leukemia Must have either anemia (hemoglobin less than 10 g/dL), thrombocytopenia (less than 100,000/mm3), cytogenetic abnormalities including +12 and 11q, elevated LDH levels, labeling index at least 2%, systemic symptoms, or hepatosplenomegaly No active CNS disease A new classification scheme for adult non-Hodgkin's lymphoma has been adopted by PDQ. The terminology of "indolent" or "aggressive" lymphoma will replace the former terminology of "low", "intermediate", or "high" grade lymphoma. However, this protocol uses the former terminology.

PATIENT CHARACTERISTICS: Age: 18 to 70 Performance status: SWOG 0-2 Life expectancy: Not specified Hematopoietic: At least 4,000/g CD34+ peripheral blood stem cells available See Disease Characteristics Hepatic: Bilirubin no greater than 1.5 mg/dL Transaminases no greater than 4 times upper limit of normal No active chronic hepatitis or liver cirrhosis Renal: Creatinine no greater than 2.0 mg/dL Cardiovascular: Left ventricular ejection fraction at least 50% Pulmonary: FEV1, FVC, and DLCO at least 50% of predicted Other: HIV negative No active infection requiring intravenous antibiotics Not pregnant or nursing Effective contraception required of all fertile patients

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: At least 4 weeks since prior chemotherapy Endocrine therapy: Prior corticosteroids allowed Radiotherapy: At least 4 weeks since prior local radiotherapy Surgery: Not specified

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 1999-01; Primary Completion 2002-12 (Actual); Study Completion 2002-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barry R. Meisenberg, MD, Study Chair — University of Maryland Greenebaum Cancer Center
Locations (1):
- Marlene & Stewart Greenebaum Cancer Center, University of Maryland, Baltimore, Maryland, United States